CLINICAL TRIAL: NCT04238169
Title: Clinical Trial Assessing the Efficacy of Abscopal Effect Induced by SBRT and Immunotherapy in Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, director physician, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-014
Record Dates: First submitted 2020-01-14; First posted 2020-01-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Non-Small-Cell Lung Cancer Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT+Toripalimab (Experimental): Immunotherapy：Toripalimab: 240 mg once every three weeks，Until progress of disease or investigators determine that clinical benefit is no longer available or there are intolerable toxicity.
  SBRT：30-50Gy/5F（2-4 locations).
  Interventions: Drug: Toripalimab; Radiation: SBRT
- SBRT+Bevacizumab+Toripalimab (Experimental): Immunotherapy：Toripalimab: 240 mg once every three weeks，Until progress of disease or investigators determine that clinical benefit is no longer available or there are intolerable toxicity.
  SBRT：30-50 Grays(Gy) in 5 fractions（2-4 locations）. Bevacizumab：7.5mg/kg once every three weeks.
  Interventions: Drug: Bevacizumab; Drug: Toripalimab; Radiation: SBRT

INTERVENTIONS:
Drug: Bevacizumab — 7.5mg/kg once every three weeks
  Arms: SBRT+Bevacizumab+Toripalimab
Drug: Toripalimab — 240 mg once every three weeks
Radiation: SBRT — 30-50Gy/5F（2-4 lesions）

SUMMARY:
This is a prospective, multicenter, open-label study to observe the effect of SBRT and immunotherapy combined with Bevacizumab or not in stage IV non-squamous non-small cell lung cancer (NSCLC) with previously failed after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Must have signed written informed consent and able to comply with study procedures.
2. Histologically and/or cytologically confirmed advanced metastatic (stage IV) non-squamous non-small cell lung cancer.
3. Previous received first-line platinum-based chemotherapy or immunotherapy (except toripalimab) and followed by progression of disease evaluated by RECIST 1.1.
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score 0-1.
6. Life expectancy ≥ 12 weeks.
7. Have at least 3 measurable lesions based on RECIST 1.1, at least 2 of them can be treated by SBRT.
8. Adequate hematologic function as defined by the following laboratory values:

   * Absolute neutrophil count ≥1.5x109/L
   * Platelets ≥80 x 109/L
   * Hemoglobin ≥9 g/dL
   * Adequate Hepatic function: Total bilirubin ≤1.5×ULN Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN OR ≤5×ULN for patients with liver metastases.
9. Adequate renal function: Creatinine ≤1.5×ULN or calculated creatinine clearance (CrCl) ≥50 mL/min and dipstick proteinuria <2+. A 24-hour urine protein test is needed if a dipstick proteinuria result of ≥2+ is detected, the proteinuria level ≤ 1g/24h.
10. International normalized ratio≤1.5 × ULN, prothrombin time (PT) or partial thromboplastin time (PTT or a PTT) ≤1.5 × ULN(within 7 days of assessment).
11. Female who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must be willing to use an adequate method of contraception.
12. Male subjects of childbearing potential must agree to use an adequate method of contraception (failure rate < 1% per year) - Contraception, starting with the first dose of study therapy through 6 months after the last dose of study therapy.

Exclusion Criteria:

1. Evidence of tumour invading major blood vessels on imaging. The investigator or the local radiologist must exclude evidence of tumour that is fully contiguous with, surrounding, or extending into the lumen of a major blood vessel (e.g., pulmonary artery or superior vena cava).
2. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device are excluded within 7 days prior to initiation of study treatment. Placement of a vascular access device should be at least 2 days prior to initiation of study treatment.
3. Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (325 mg/day) or other nonsteroidal anti-inflammatory agents known to inhibit platelet function.
4. Current or recent (within 10 days of first dose of bevacizumab) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes. Prophylactic use of anticoagulants is allowed.
5. History or evidence of inherited bleeding diathesis or coagulopathy that increases the risk of bleeding.
6. Uncontrolled hypertension (blood pressures: systolic>150 mmHg and/or diastolic >100 mmHg).

   Prior history of hypertensive crisis or hypertensive encephalopathy.
7. Clinically significant (i.e., active) cardiovascular disease, including but not limited to cerebral vascular accident (CVA) or (transient ischemic attack) TIA (≤6 months before randomization), myocardial infarction (≤6 months before randomization), unstable angina, congestive heart failure New York Heart Association Class≥II, or serious cardiac arrhythmia requiring medication during the study and that might interfere with regularity of the study treatment or not controlled by medication.
8. Significant vascular disease (including but not limited to aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization.
9. The lesion has received prior radiotherapy and is not suitable for SBRT.
10. Has stable brain metastases is allowed, but the brain metastases will not receive SBRT or whole brain radiotherapy (WBRT)
11. Malignancies other than NSCLC within 2 years except for basal or squamous cell skin cancer, carcinoma in situ of the cervix and cured early stage prostate cancer.
12. Corticosteroid therapy at a dose equivalent to 10 mg prednisone per day or any other systemic immunosuppressive therapy within 14 days prior to randomization. Topical or inhaled steroids are permitted. Taking immunosuppressive drugs accidentally during the trial will be allowed, but it is strongly recommended to reduce the dose as soon as possible.
13. A positive HIV test result, presence of active HIV, hepatitis B or hepatitis C（evaluate at local laboratories）
14. Non-healing wound, active peptic ulcer, or bone fracture.
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of enrollment.
16. Pregnant or lactating, or intending to become pregnant during the study.
17. Treatment with any other investigational agent or participation in another clinical trial within 28 days prior to randomization.
18. Evidence of ongoing or active infection requiring IV antibiotics; any other disease, neurological, or metabolic dysfunction; physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
19. Patients diagnosed with a tracheo-oesophageal fistula.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 6 months
  Assess the efficacy (overall response rate [ORR]) of SBRT and Toripalimab combined with Bevacizumab or not in stage IV non-squamous NSCLC with previously failed after chemotherapy. (according to RECIST version 1.1 and EORTC 1999)
Objective response of non-target lesion | Up to 6 months
  Assess the efficacy (Objective response of non-target lesion) of SBRT and Toripalimab combined with Bevacizumab or not in stage IV non-squamous NSCLC with previously failed after chemotherapy. (according to RECIST version 1.1 and EORTC 1999)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  Estimate the progression-free survival (PFS) in patients with NSCLC
Duration of response | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Overall survival | From date of first dose of study drug until withdrawal of consent or death (up to approximately 2 years)
  Duration from the date of initial treatment to the date of death due to any cause.
The incidence of adverse events (AEs) as a measure of safety | For each participant, from the first participant first dose until 30 days after the last dose (up to approximately 2 years)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered an investigational product. Safety and tolerance evaluated by incidence, severity and outcomes of AEs (according to NCI-CTCAE 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality, China